CLINICAL TRIAL: NCT05114369
Title: Does Timing of Completion Radical Cholecystectomy Determine the Survival Outcome in Incidental Carcinoma Gallbladder - a Single Center Retrospective Analysis
Brief Title: Does Timing of Completion Radical Cholecystectomy Determine the Survival in Incidental Carcinoma Gallbladder
Acronym: IGBC
Status: Completed | Type: Observational
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Sponsor
Other Study IDs: 00
Record Dates: First submitted 2021-10-11; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Gall Bladder Carcinoma; Survival
Keywords: Incidental; Gallbladder cancer; Re-resection; Survival
MeSH Terms: conditions — Gallbladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Early (<4weeks), Intermediate (4-12 weeks) and Late (>12 weeks): Interval between index cholecystectomy and radical re-resection with curative intent
  Interventions: Procedure: Curative surgery

INTERVENTIONS:
Procedure: Curative surgery

SUMMARY:
Various factors determine the long term survival in this non-uniform cohort of incidental gallbladder cancer. Timing of re-intervention is suggested to play an important role in the outcome. Few centers are proponents of early surgery in order to prevent dissemination, while others have suggested an intentional delay of 3 months to filter out cases with aggressive pathology. In the present study, investigators intend to evaluate the factors affecting survival in incidental Gallbladder Cancer (IGBC) with special reference to timing of re-intervention.

DETAILED DESCRIPTION:
Surgical Gastroenterology department at our institute is a tertiary referral center for hepatobiliary malignancies; covering a large part of North and North-east India. The details and progress reports of patients of Gallbladder Cancer (GBC) being referred to and treated at the institute is maintained in a prospective manner on hospital data base. This includes demographic data, presenting complains, details of relevant investigations done outside and in the hospital, previous surgery, pre-hospital course, operative findings, post operative course and final histopathology. Being a retrospective analysis of data not affecting clinical outcomes, ethical approval was not taken. During the study period (Jan 2009 to Dec 2018), 1049 participants with diagnosis of GBC (including 91 IGBC participants) were admitted; 239/958 participants with diagnosis of GBC and 48/91 with diagnosis of GBC could undergo resection with curative intent. Information regarding adjuvant therapy, recurrence, and survival were retrieved through data maintained on follow up out-patient cards till December 2019. Few participants who stopped visiting the hospital were contacted telephonically or through letters. All available histopathology blocks and slides following the index cholecystectomy were re-reviewed by the pathologists in the institute. Tumor type, differentiation and primary T stage were documented for majority of cases. Interval between index cholecystectomy and date of re-operation was calculated for all the participants and divided into 3 groups: Early (<4weeks), Intermediate (4-12 weeks) and Late (>12 weeks). Primary objective was to assess the effect of tumor characteristics and the time gap (between index surgery and re-resection) on overall survival following curative (R0/R1) resection.

ELIGIBILITY:
Inclusion Criteria:

All incidental carcinoma gallbladder patients who could undergo curative resection during the study period (Jan 2009 to Dec 2018)

Exclusion Criteria:

Metastasis on preoperative investigation or on staging laparoscopy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All incidental carcinoma gallbladder patients who were admitted for possible curative resection during the study period (Jan 2009 to Dec 2018)
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Survival based on timing of completion radical cholecystectomy | 01.01.2009 to 31.12.2018
  Overall and disease free survival

SECONDARY OUTCOMES:
Determinants of factors associated with survival in incidental gallbladder carcinoma | 01.01.2009 to 31.12.2018
  Factors related to primary surgery (residual disease, primary T stage), type of resection (Wedge resection, Segment 4B-5 excision or Common bile duct excision), tumor characteristics (differentiation and lymohovascular invasion) and final stage (AJCC 8th edition)

IPD SHARING:
Plan to Share IPD: No
The final data sheet can be shared and not the individual data as the data was retrieved from online database

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT05114369/Prot_SAP_000.pdf